CLINICAL TRIAL: NCT00262340
Title: Prospective, Randomised Controlled Trial of the Use of Inflammatory Markers to Guide Therapy in Children With Severe Asthma
Brief Title: The Use of Inflammatory Markers to Guide Therapy in Children With Severe Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: National Heart and Lung Institute (Other); Imperial College London (Other); British Lung Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05/Q0404/30
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
Keywords: Asthma; Pediatrics; Airway; Inflammation
MeSH Terms: conditions — Asthma; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): This arm will have treatment changed based on measures of inflammation
  Interventions: Other: Non invasive measurement of airway inflammation
- 2 (Active Comparator): Treatment will be changed on the basis of reported asthma symptoms
  Interventions: Other: Non invasive measurement of airway inflammation

INTERVENTIONS:
Other: Non invasive measurement of airway inflammation — Airway inflammation will be assessed non-invasively using induced sputum and exhaled nitric oxide. In the active group the results of these tests will be used to determine if asthma treatment should be changed. In the comparator group treatment changes will be based according to conventional symptom based management

SUMMARY:
The purpose of this study is to determine whether using non-invasive measurements of airway inflammation can improve clinical decision making in children with severe asthma compared to conventional management (British Thoracic Society Guidelines)

DETAILED DESCRIPTION:
Children with severe asthma pose a management dilemma; it is difficult to reduce their treatment while they are symptomatic, but the plateau of the dose response curve for inhaled corticosteroids (ICS) may have been reached. Studies in symptomatic adults and asymptomatic children with asthma suggest measuring induced sputum eosinophils allows better asthma management. We will recruit 80 children with severe asthma (treated with at least 500 mcg/day inhaled fluticasone or equivalent). We will see them every three months for a year, and perform sputum induction and measurements of exhaled nitric oxide (eNO). Half will be randomised to conventional management; half will have a reduction of ICS if there are no sputum eosinophils, or (if a sample cannot be produced) eNO is normal. The trial endpoint is whether there is a significant reduction in the median dose of ICS in the inflammatory markers group, with no increase in total number of asthma exacerbations. This study is also hypothesis generating. We will use our panel of markers (a) to try to improve clinical monitoring; and (b) to determine the molecular mechanisms of relapse of severe asthma.

ELIGIBILITY:
Inclusion Criteria:

Children >8 years with severe asthma defined as:

Taking at least 500mcg fluticasone propionate (or equivalent) per day, plus a long acting beta agonist plus a leukotriene antagonist or previous trial

Exclusion Criteria:

Children taking steroid sparing agent (cyclosporin, azathioprine, methotrexate) Children with other major respiratory diagnoses such as bronchiectasis

-

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2005-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Number of exacerbations; | 1 year
Number of symptom free days and bronchodilator use per week | 1 year

SECONDARY OUTCOMES:
Doses of inhaled and oral corticosteroid used per year | 1 year
Comparison of daily versus single visit measures of eNO to predict an asthma exacerbation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bush, MBBS, Principal Investigator — Imperial College of Science Technology and Medicine, National Heart and Lung Institue
Locations (1):
- Royal Brompton Hospital, London, United Kingdom